CLINICAL TRIAL: NCT04014283
Title: Prevention of Females Malignancies in Families With Hereditary Breast Cancer by Personalized Optimization of Se Levels in the Organism.
Brief Title: Prevention of Female Cancers by Optimization of Selenium Levels in the Organism.
Acronym: SELINA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Read-Gene S.A. (Other)
Collaborators: National Center for Research and Development, Poland (Other); IQ Pharma S.A. (Unknown); West Pomeranian University of Technology (Unknown); Vipharm S.A. (Unknown)
Responsible Party: Principal Investigator, Lubinski Jan, MD, PhD, Read-Gene S.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INNOMED/I/16?NCBR/2014
Record Dates: First submitted 2019-06-18; First posted 2019-07-10 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Breast Neoplasms
Keywords: Selenium; Supplement; Prevention; Females; Risk
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Supplementation of selenium or diet modification will be effective in reducing the risk of developing breast cancer in women with high risk, as compared to placebo.
  The null hypothesis assumes no significant differences between the supplementation and placebo groups. The alternative hypothesis assumes that patients with high risk of breast cancer in supplementation or diet modification group with optimal selenium level will have significantly reduced risk of developing cancer in relation to the placebo group with selenium deficiency. The comparison of disease-free survival time intervals is best covered by Cox Regression and is represented by a Kaplan-Meier survival curve tested by log- rank test.
  The comparison of proportions of diseased and healthy subjects in the supplementation arm with respect to the placebo arm is best attempted using the Fisher Exact Test. Graphical representation should be based on bar plots for percentages and/or raw numbers, or a similar representation.
Who Masked: Investigator
Masking Description: The selected randomization method is block randomization with randomly chosen blocks sizes.
  Randomization must take place before 120 days after the Screening Visit (Day 0). After confirmation that the patient meets all eligibility criteria for the study, the patient will be randomly assigned (1:1) to either placebo or supplementation group. Patients with selenium deficiency can choose between diet modification and supplementation group.
  The last step of randomisation is the blinding/assigning procedure - connecting randomization numbers with placebo or supplement packages numbers and assigning them to the subjects. All SELINA personnel, participants and clinicians will be blinded to the treatment allocation; only the Statistical Center will have the possibility to unblind the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BRCA(+) Selenium deficiency (Active Comparator): Placebo: 100 Supplement: 100
  Interventions: Dietary Supplement: Selenium supplementation or placebo treatment
- BRCA(+) Selenium excess (Active Comparator): Diet modification: 500 Observation: 500
  Interventions: Other: Diet modification
- BRCA(-) Selenium deficiency (Active Comparator): Placebo: 900 Supplement: 900 Diet modification: 900 Observation: 900
  Interventions: Other: Selenium supplementation or placebo treatment and diet modification
- BRCA(-) Selenium excess (Active Comparator): Diet modification: 1100 Observation: 1100
  Interventions: Other: Diet modification
- BRCA(+) Selenium excess, age > 50 (Active Comparator): Diet modification: 200 Observation: 200
  Interventions: Other: Diet modification

INTERVENTIONS:
Dietary Supplement: Selenium supplementation or placebo treatment — Patients from this group will receive selenium supplement to achieve optimal selenium level
  Arms: BRCA(+) Selenium deficiency
Other: Diet modification — Patients from this group will have modified diet over the course of the study. Diet modification is aimed to lower selenium concentration in blood.
  Arms: BRCA(+) Selenium excess; BRCA(+) Selenium excess, age > 50; BRCA(-) Selenium excess
Other: Selenium supplementation or placebo treatment and diet modification — In this group patients will receive supplement, placebo or diet modification. The goal is to raise selenium concentration in blood
  Arms: BRCA(-) Selenium deficiency

SUMMARY:
Hypothesis to be tested:

Oral supplementation or diet modifications of selenium to a specified range will be effective in reducing the risk of developing cancer of any type in women with high risk of breast cancer, as compared to placebo.

DETAILED DESCRIPTION:
Primary Objective

• To determine the efficacy of oral daily supplementation or diet modification of selenium to an optimal level compared to placebo, in reducing the incidence of any cancers in an at risk population of women over the 60 months of the study.

Secondary Objectives

* To determine the efficacy of oral daily supplementation or diet modification of selenium to an optimal level compared to placebo, in reducing the incidence of breast cancer in an at risk population of women over the 60 months of the study.
* To explore the relationship between the effects of study supplement or diet modifications on cancer risk and genetic factors.

The study will have 7000 participants. All the measurements will be performed via blood tests.

ELIGIBILITY:
Inclusion Criteria:

- Sub-group I - BRCA1 mutation carriers

1. Carrier-status of BRCA1 mutation
2. Age >20 years
3. Have a breast magnetic resonance imaging and/or ultrasonography and/or mammography that reveals no disease at maximum 9 months after enrollment
4. Be able to give information consent and sign an informed consent form
5. Be willing to comply with all of the study procedures as per the protocol
6. Be willing to inform researchers about current or any new pregnancy
7. Sub-optimal Se level in the blood

Sub-group II - Females from families with hereditary breast cancers but without BRCA1 mutations

1. Age ≥40 years
2. Age ≥20 years for women that have been diagnosed previously with breast cancer
3. Positive medical history of family, matching criteria of hereditary breast/ovarian cancer (HBO) (Appendix 1)
4. No personal history of cancer except for breast cancer and non-melanoma skin cancers
5. Have a breast magnetic resonance imaging/ultrasonography/mammography that reveals no disease at maximum 9 months after enrollment
6. Be able to give information consent and sign an informed consent form
7. Absence of BRCA1 mutations after testing for at least three founder mutations (BRCA1 5382insC, BRCA1 300T/G, BRCA1 4154delA)
8. Be willing to comply with all of the study procedures as per the protocol
9. Be willing to inform researchers about current or any new pregnancy
10. Sub-optimal Se level in the blood

Exclusion Criteria:

Sub-group I - BRCA1 mutation carriers

1. Diagnosis of any previous cancer except for breast cancers and non-melanoma skin cancers
2. Absence of a magnetic resonance imaging/ultrasonography/mammography that reveals no disease at maximum 9 months after enrollment
3. Current pregnancy or breast-feeding
4. Optimal Se level in the blood
5. Age <20 years
6. Any medical illness, which, in the investigator's opinion, cannot be adequately controlled with appropriate therapy
7. Participation in any other clinical study involving a medical, surgical, nutritional, or life-style intervention (unless individuals are no longer receiving any intervention and they are in the follow-up phase only)

Sub-group II - Females from families with hereditary breast cancers but without BRCA1 mutations

1. Diagnosis of any previous cancer except for breast cancers and non-melanoma skin cancers
2. Absence of magnetic resonance imaging and/or ultrasonography and/or mammography that reveals no disease at maximum 9 months after enrollment
3. Absence of matching pedigree/clinical/molecular criteria of HBO (Appendix 1)
4. Presence of BRCA1 mutation
5. Current pregnancy or breast-feeding
6. Optimal Se level in the blood
7. Age <40 years except for women that have been previously diagnosed with breast cancer
8. Any medical illness, which, in the investigator's opinion, cannot be adequately controlled with appropriate therapy
9. Participation in any other clinical study involving a medical, surgical, nutritional, or life-style intervention (unless individuals are no longer receiving any intervention and they are in the follow-up phase only)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Development of any new cancer | within 60 months of the study
  Cancer diagnosis will be determined by routine clinical management and confirmed by central pathology review. Cancer-free survival is defined as the period of time between randomization and diagnosis of cancer, or - for patients who do not develop cancer - the period of time between randomization and last contact or death unrelated to cancer.

SECONDARY OUTCOMES:
Development of new breast cancer | within 60 months of the study
  Cancer diagnosis will be determined by routine clinical management and confirmed by central pathology review. Cancer-free survival is defined as the period of time between randomization and diagnosis of cancer, or - for patients who do not develop cancer - the period of time between randomization and last contact or death unrelated to cancer.
Proportion of any other cancers (besides breast cancers) at the end of 60 months | within 60 months of the study
  Cancer diagnosis will be determined by routine clinical management and confirmed by central pathology review. Cancer-free survival is defined as the period of time between randomization and diagnosis of cancer, or - for patients who do not develop cancer - the period of time between randomization and last contact or death unrelated to cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Lubiński, MD, PhD, Principal Investigator — Read-Gene S.A.; Cezary Cybulski, MD, PhD, Study Chair — Read-Gene S.A.; Jacek Gronwald, MD, PhD, Study Chair — Read-Gene S.A.; Tomasz Huzarski, MD, PhD, Study Chair — Read-Gene S.A.; Anna Jakubowska, MD, PhD, Study Chair; Antoni Morawski, PhD, Study Chair; Ewa Stachowska, PhD, Study Chair — Read-Gene S.A.; Edyta Balejko, PhD, Study Chair; Karolina Ertmańska, PhD, Study Chair
Locations (1):
- Read-Gene S.A., Grzepnica, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
We still did not collect all the required participants. It is hard to tell that the data could be useful later on.

REFERENCES:
- [Background] Adeoti ML, Oguntola AS, Akanni EO, Agodirin OS, Oyeyemi GM. Trace elements; copper, zinc and selenium, in breast cancer afflicted female patients in LAUTECH Osogbo, Nigeria. Indian J Cancer. 2015 Jan-Mar;52(1):106-9. doi: 10.4103/0019-509X.175573. PMID 26837992
- [Background] Algotar AM, Behnejad R, Singh P, Thompson PA, Hsu CH, Stratton SP. EFFECT OF SELENIUM SUPPLEMENTATION ON PROTEOMIC SERUM BIOMARKERS IN ELDERLY MEN. J Frailty Aging. 2015;4(2):107-10. doi: 10.14283/jfa.2015.48. PMID 26366377
- [Background] Arnaud J, Arnault N, Roussel AM, Bertrais S, Ruffieux D, Galan P, Favier A, Hercberg S. Relationships between selenium, lipids, iron status and hormonal therapy in women of the SU.VI.M.AX cohort. J Trace Elem Med Biol. 2007;21 Suppl 1:66-9. doi: 10.1016/j.jtemb.2007.09.025. Epub 2007 Oct 22. PMID 18039502
- [Background] Barany E, Bergdahl IA, Bratteby LE, Lundh T, Samuelson G, Skerfving S, Oskarsson A. Iron status influences trace element levels in human blood and serum. Environ Res. 2005 Jun;98(2):215-23. doi: 10.1016/j.envres.2004.09.010. PMID 15820728
- [Background] Singh BP, Dwivedi S, Dhakad U, Murthy RC, Choubey VK, Goel A, Sankhwar SN. Status and Interrelationship of Zinc, Copper, Iron, Calcium and Selenium in Prostate Cancer. Indian J Clin Biochem. 2016 Mar;31(1):50-6. doi: 10.1007/s12291-015-0497-x. Epub 2015 Apr 16. PMID 26855488
- [Background] Bleys J, Navas-Acien A, Guallar E. Serum selenium levels and all-cause, cancer, and cardiovascular mortality among US adults. Arch Intern Med. 2008 Feb 25;168(4):404-10. doi: 10.1001/archinternmed.2007.74. PMID 18299496
- [Background] Borawska MH, Socha K, Lazarczyk B, Czyzewska E, Markiewicz R, Darewicz B. The effects of diet on selenium concentration in serum in patients with cancer. Nutr Cancer. 2009;61(5):629-33. doi: 10.1080/01635580902825555. PMID 19838936
- [Background] Chareonpong-Kawamoto N, Yasumoto K. Selenium deficiency as a cause of overload of iron and unbalanced distribution of other minerals. Biosci Biotechnol Biochem. 1995 Feb;59(2):302-6. doi: 10.1271/bbb.59.302. PMID 7766029
- [Background] Chmielnicka J, Zareba G, Witasik M, Brzeznicka E. Zinc-selenium interaction in the rat. Biol Trace Elem Res. 1988 Jan-Apr;15:267-76. doi: 10.1007/BF02990143. PMID 2484524
- [Background] Clark LC, Combs GF Jr, Turnbull BW, Slate EH, Chalker DK, Chow J, Davis LS, Glover RA, Graham GF, Gross EG, Krongrad A, Lesher JL Jr, Park HK, Sanders BB Jr, Smith CL, Taylor JR. Effects of selenium supplementation for cancer prevention in patients with carcinoma of the skin. A randomized controlled trial. Nutritional Prevention of Cancer Study Group. JAMA. 1996 Dec 25;276(24):1957-63. PMID 8971064
- [Background] Coates RJ, Weiss NS, Daling JR, Morris JS, Labbe RF. Serum levels of selenium and retinol and the subsequent risk of cancer. Am J Epidemiol. 1988 Sep;128(3):515-23. doi: 10.1093/oxfordjournals.aje.a114999. PMID 3046338
- [Background] Combs GF Jr, Gray WP. Chemopreventive agents: selenium. Pharmacol Ther. 1998 Sep;79(3):179-92. doi: 10.1016/s0163-7258(98)00014-x. PMID 9776375
- [Background] Combs GF Jr, Clark LC, Turnbull BW. An analysis of cancer prevention by selenium. Biofactors. 2001;14(1-4):153-9. doi: 10.1002/biof.5520140120. PMID 11568452
- [Background] Constantinescu S, Hecht K, Sobotzki N, Erzinger MM, Bovet C, Shay JW, Wollscheid B, Sturla SJ, Marra G, Beerenwinkel N. Transcriptomic responses of cancerous and noncancerous human colon cells to sulforaphane and selenium. Chem Res Toxicol. 2014 Mar 17;27(3):377-86. doi: 10.1021/tx400427t. Epub 2014 Jan 13. PMID 24383545
- [Background] Druesne-Pecollo N, Touvier M, Barrandon E, Chan DS, Norat T, Zelek L, Hercberg S, Latino-Martel P. Excess body weight and second primary cancer risk after breast cancer: a systematic review and meta-analysis of prospective studies. Breast Cancer Res Treat. 2012 Oct;135(3):647-54. doi: 10.1007/s10549-012-2187-1. Epub 2012 Aug 5. PMID 22864804
- [Background] Duffield-Lillico AJ, Dalkin BL, Reid ME, Turnbull BW, Slate EH, Jacobs ET, Marshall JR, Clark LC; Nutritional Prevention of Cancer Study Group. Selenium supplementation, baseline plasma selenium status and incidence of prostate cancer: an analysis of the complete treatment period of the Nutritional Prevention of Cancer Trial. BJU Int. 2003 May;91(7):608-12. doi: 10.1046/j.1464-410x.2003.04167.x. PMID 12699469
- [Background] Duffield-Lillico AJ, Reid ME, Turnbull BW, Combs GF Jr, Slate EH, Fischbach LA, Marshall JR, Clark LC. Baseline characteristics and the effect of selenium supplementation on cancer incidence in a randomized clinical trial: a summary report of the Nutritional Prevention of Cancer Trial. Cancer Epidemiol Biomarkers Prev. 2002 Jul;11(7):630-9. PMID 12101110
- [Background] El-Bayoumy K, Das A, Russell S, Wolfe S, Jordan R, Renganathan K, Loughran TP, Somiari R. The effect of selenium enrichment on baker's yeast proteome. J Proteomics. 2012 Jan 4;75(3):1018-30. doi: 10.1016/j.jprot.2011.10.013. Epub 2011 Oct 29. PMID 22067702
- [Background] Garland M, Morris JS, Stampfer MJ, Colditz GA, Spate VL, Baskett CK, Rosner B, Speizer FE, Willett WC, Hunter DJ. Prospective study of toenail selenium levels and cancer among women. J Natl Cancer Inst. 1995 Apr 5;87(7):497-505. doi: 10.1093/jnci/87.7.497. PMID 7707436
- [Background] Geybels MS, van den Brandt PA, Schouten LJ, van Schooten FJ, van Breda SG, Rayman MP, Green FR, Verhage BA. Selenoprotein gene variants, toenail selenium levels, and risk for advanced prostate cancer. J Natl Cancer Inst. 2014 Mar;106(3):dju003. doi: 10.1093/jnci/dju003. Epub 2014 Feb 22. PMID 24563517
- [Background] Geybels MS, Hutter CM, Kwon EM, Ostrander EA, Fu R, Feng Z, Stanford JL, Peters U. Variation in selenoenzyme genes and prostate cancer risk and survival. Prostate. 2013 May;73(7):734-42. doi: 10.1002/pros.22617. Epub 2012 Nov 9. PMID 23143801
- [Background] Ha EJ, Smith AM. Plasma selenium and plasma and erythrocyte glutathione peroxidase activity increase with estrogen during the menstrual cycle. J Am Coll Nutr. 2003 Feb;22(1):43-51. doi: 10.1080/07315724.2003.10719274. PMID 12569113
- [Background] Hortobagyi GN, de la Garza Salazar J, Pritchard K, Amadori D, Haidinger R, Hudis CA, Khaled H, Liu MC, Martin M, Namer M, O'Shaughnessy JA, Shen ZZ, Albain KS; ABREAST Investigators. The global breast cancer burden: variations in epidemiology and survival. Clin Breast Cancer. 2005 Dec;6(5):391-401. doi: 10.3816/cbc.2005.n.043. PMID 16381622
- [Background] Jablonska E, Gromadzinska J, Sobala W, Reszka E, Wasowicz W. Lung cancer risk associated with selenium status is modified in smoking individuals by Sep15 polymorphism. Eur J Nutr. 2008 Feb;47(1):47-54. doi: 10.1007/s00394-008-0696-9. Epub 2008 Jan 31. PMID 18239845
- [Background] Johnson CC, Fordyce FM, Rayman MP. Symposium on 'Geographical and geological influences on nutrition': Factors controlling the distribution of selenium in the environment and their impact on health and nutrition. Proc Nutr Soc. 2010 Feb;69(1):119-32. doi: 10.1017/S0029665109991807. Epub 2009 Dec 8. PMID 19968907
- [Background] Kim JH, Hue JJ, Kang BS, Park H, Nam SY, Yun YW, Kim JS, Lee BJ. Effects of selenium on colon carcinogenesis induced by azoxymethane and dextran sodium sulfate in mouse model with high-iron diet. Lab Anim Res. 2011 Mar;27(1):9-18. doi: 10.5625/lar.2011.27.1.9. Epub 2011 Mar 25. PMID 21826154
- [Background] Klein EA, Thompson IM Jr, Tangen CM, Crowley JJ, Lucia MS, Goodman PJ, Minasian LM, Ford LG, Parnes HL, Gaziano JM, Karp DD, Lieber MM, Walther PJ, Klotz L, Parsons JK, Chin JL, Darke AK, Lippman SM, Goodman GE, Meyskens FL Jr, Baker LH. Vitamin E and the risk of prostate cancer: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2011 Oct 12;306(14):1549-56. doi: 10.1001/jama.2011.1437. PMID 21990298
- [Background] Knekt P, Marniemi J, Teppo L, Heliovaara M, Aromaa A. Is low selenium status a risk factor for lung cancer? Am J Epidemiol. 1998 Nov 15;148(10):975-82. doi: 10.1093/oxfordjournals.aje.a009574. PMID 9829869
- [Background] Kristal AR, Darke AK, Morris JS, Tangen CM, Goodman PJ, Thompson IM, Meyskens FL Jr, Goodman GE, Minasian LM, Parnes HL, Lippman SM, Klein EA. Baseline selenium status and effects of selenium and vitamin e supplementation on prostate cancer risk. J Natl Cancer Inst. 2014 Mar;106(3):djt456. doi: 10.1093/jnci/djt456. Epub 2014 Feb 22. PMID 24563519
- [Background] Laclaustra M, Stranges S, Navas-Acien A, Ordovas JM, Guallar E. Serum selenium and serum lipids in US adults: National Health and Nutrition Examination Survey (NHANES) 2003-2004. Atherosclerosis. 2010 Jun;210(2):643-8. doi: 10.1016/j.atherosclerosis.2010.01.005. Epub 2010 Jan 11. PMID 20102763
- [Background] Lippman SM, Klein EA, Goodman PJ, Lucia MS, Thompson IM, Ford LG, Parnes HL, Minasian LM, Gaziano JM, Hartline JA, Parsons JK, Bearden JD 3rd, Crawford ED, Goodman GE, Claudio J, Winquist E, Cook ED, Karp DD, Walther P, Lieber MM, Kristal AR, Darke AK, Arnold KB, Ganz PA, Santella RM, Albanes D, Taylor PR, Probstfield JL, Jagpal TJ, Crowley JJ, Meyskens FL Jr, Baker LH, Coltman CA Jr. Effect of selenium and vitamin E on risk of prostate cancer and other cancers: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2009 Jan 7;301(1):39-51. doi: 10.1001/jama.2008.864. Epub 2008 Dec 9. PMID 19066370
- [Background] Lubiński J. (red.), Genetyka Kliniczna Nowotworów 2015; ISBN 978-83-61350-95-8
- [Background] Maciel-Dominguez A, Swan D, Ford D, Hesketh J. Selenium alters miRNA profile in an intestinal cell line: evidence that miR-185 regulates expression of GPX2 and SEPSH2. Mol Nutr Food Res. 2013 Dec;57(12):2195-205. doi: 10.1002/mnfr.201300168. Epub 2013 Aug 12. PMID 23934683
- [Background] Mark SD, Qiao YL, Dawsey SM, Wu YP, Katki H, Gunter EW, Fraumeni JF Jr, Blot WJ, Dong ZW, Taylor PR. Prospective study of serum selenium levels and incident esophageal and gastric cancers. J Natl Cancer Inst. 2000 Nov 1;92(21):1753-63. doi: 10.1093/jnci/92.21.1753. PMID 11058618
- [Background] Martinez EE, Darke AK, Tangen CM, Goodman PJ, Fowke JH, Klein EA, Abdulkadir SA. A functional variant in NKX3.1 associated with prostate cancer risk in the Selenium and Vitamin E Cancer Prevention Trial (SELECT). Cancer Prev Res (Phila). 2014 Sep;7(9):950-7. doi: 10.1158/1940-6207.CAPR-14-0075. Epub 2014 Jun 3. PMID 24894197
- [Background] Massafra C, Gioia D, De Felice C, Picciolini E, De Leo V, Bonifazi M, Bernabei A. Effects of estrogens and androgens on erythrocyte antioxidant superoxide dismutase, catalase and glutathione peroxidase activities during the menstrual cycle. J Endocrinol. 2000 Dec;167(3):447-52. doi: 10.1677/joe.0.1670447. PMID 11115771
- [Background] Narod SA. BRCA mutations in the management of breast cancer: the state of the art. Nat Rev Clin Oncol. 2010 Dec;7(12):702-7. doi: 10.1038/nrclinonc.2010.166. Epub 2010 Oct 19. PMID 20956982
- [Background] Okuno T, Miura K, Sakazaki F, Nakamuro K, Ueno H. Methylseleninic acid (MSA) inhibits 17beta-estradiol-induced cell growth in breast cancer T47D cells via enhancement of the antioxidative thioredoxin/ thioredoxin reductase system. Biomed Res. 2012;33(4):201-10. doi: 10.2220/biomedres.33.201. PMID 22975630
- [Background] Penney KL, Schumacher FR, Li H, Kraft P, Morris JS, Kurth T, Mucci LA, Hunter DJ, Kantoff PW, Stampfer MJ, Ma J. A large prospective study of SEP15 genetic variation, interaction with plasma selenium levels, and prostate cancer risk and survival. Cancer Prev Res (Phila). 2010 May;3(5):604-10. doi: 10.1158/1940-6207.CAPR-09-0216. Epub 2010 Apr 27. PMID 20424130
- [Background] Peters U, Takata Y. Selenium and the prevention of prostate and colorectal cancer. Mol Nutr Food Res. 2008 Nov;52(11):1261-72. doi: 10.1002/mnfr.200800103. PMID 18763256
- [Background] Petkova-Marinova T, B Ruseva, B Atanasova, B Paneva-Barzashka, P Laleva and V Petrov; Relationships between parameters of iron metabolism and serum concentrations of copper and selenium in women with normal and problem pregnancies; Merit Research Journal of Medicine and Medical Sciences (ISSN: 2354-323X) Vol. 4(8) pp. 406-414, August, 2016
- [Background] Polish Ministry of Health, Programme for diagnostics and management of families with hereditary predisposition to breast and ovarian cancers
- [Background] Pourmand G, Salem S, Moradi K, Nikoobakht MR, Tajik P, Mehrsai A. Serum selenium level and prostate cancer: a case-control study. Nutr Cancer. 2008;60(2):171-6. doi: 10.1080/01635580701627277. PMID 18444148
- [Background] Rayman MP. Selenium and human health. Lancet. 2012 Mar 31;379(9822):1256-68. doi: 10.1016/S0140-6736(11)61452-9. Epub 2012 Feb 29. PMID 22381456
- [Background] Rayman MP. Selenium in cancer prevention: a review of the evidence and mechanism of action. Proc Nutr Soc. 2005 Nov;64(4):527-42. doi: 10.1079/pns2005467. PMID 16313696
- [Background] Reid ME, Duffield-Lillico AJ, Garland L, Turnbull BW, Clark LC, Marshall JR. Selenium supplementation and lung cancer incidence: an update of the nutritional prevention of cancer trial. Cancer Epidemiol Biomarkers Prev. 2002 Nov;11(11):1285-91. PMID 12433704
- [Background] Reid ME, Duffield-Lillico AJ, Sunga A, Fakih M, Alberts DS, Marshall JR. Selenium supplementation and colorectal adenomas: an analysis of the nutritional prevention of cancer trial. Int J Cancer. 2006 Apr 1;118(7):1777-81. doi: 10.1002/ijc.21529. PMID 16217756
- [Background] Robson M, Offit K. Clinical practice. Management of an inherited predisposition to breast cancer. N Engl J Med. 2007 Jul 12;357(2):154-62. doi: 10.1056/NEJMcp071286. No abstract available. PMID 17625127
- [Background] Sandstrom B. Micronutrient interactions: effects on absorption and bioavailability. Br J Nutr. 2001 May;85 Suppl 2:S181-5. PMID 11509108
- [Background] Schrauzer GN. Selenomethionine: a review of its nutritional significance, metabolism and toxicity. J Nutr. 2000 Jul;130(7):1653-6. doi: 10.1093/jn/130.7.1653. PMID 10867031
- [Background] Schrauzer GN, White DA, Schneider CJ. Cancer mortality correlation studies--III: statistical associations with dietary selenium intakes. Bioinorg Chem. 1977;7(1):23-31. doi: 10.1016/s0006-3061(00)80126-x. PMID 856291
- [Background] Semba RD, Ricks MO, Ferrucci L, Xue QL, Guralnik JM, Fried LP. Low serum selenium is associated with anemia among older adults in the United States. Eur J Clin Nutr. 2009 Jan;63(1):93-9. doi: 10.1038/sj.ejcn.1602889. Epub 2007 Sep 5. PMID 17805227
- [Background] Shah YM, Kaul A, Dong Y, Ip C, Rowan BG. Attenuation of estrogen receptor alpha (ERalpha) signaling by selenium in breast cancer cells via downregulation of ERalpha gene expression. Breast Cancer Res Treat. 2005 Aug;92(3):239-50. doi: 10.1007/s10549-005-3203-5. PMID 16155795
- [Background] Slattery ML, Lundgreen A, Welbourn B, Corcoran C, Wolff RK. Genetic variation in selenoprotein genes, lifestyle, and risk of colon and rectal cancer. PLoS One. 2012;7(5):e37312. doi: 10.1371/journal.pone.0037312. Epub 2012 May 17. PMID 22615972
- [Background] Smith AM, Chang MP, Medeiros LC. Generational differences in selenium status of women. Biol Trace Elem Res. 2000 Summer;75(1-3):157-65. doi: 10.1385/BTER:75:1-3:157. PMID 11051605
- [Background] Speckmann B, Grune T. Epigenetic effects of selenium and their implications for health. Epigenetics. 2015;10(3):179-90. doi: 10.1080/15592294.2015.1013792. PMID 25647085
- [Background] Steinbrecher A, Meplan C, Hesketh J, Schomburg L, Endermann T, Jansen E, Akesson B, Rohrmann S, Linseisen J. Effects of selenium status and polymorphisms in selenoprotein genes on prostate cancer risk in a prospective study of European men. Cancer Epidemiol Biomarkers Prev. 2010 Nov;19(11):2958-68. doi: 10.1158/1055-9965.EPI-10-0364. Epub 2010 Sep 17. PMID 20852007
- [Background] van den Brandt PA, Goldbohm RA, van't Veer P, Bode P, Dorant E, Hermus RJ, Sturmans F. Toenail selenium levels and the risk of breast cancer. Am J Epidemiol. 1994 Jul 1;140(1):20-6. doi: 10.1093/oxfordjournals.aje.a117155. PMID 8017400
- [Background] van den Brandt PA, Goldbohm RA, van 't Veer P, Bode P, Dorant E, Hermus RJ, Sturmans F. A prospective cohort study on selenium status and the risk of lung cancer. Cancer Res. 1993 Oct 15;53(20):4860-5. PMID 8402674
- [Background] van Noord PA, Maas MJ, van der Tweel I, Collette C. Selenium and the risk of postmenopausal breast cancer in the DOM cohort. Breast Cancer Res Treat. 1993;25(1):11-9. doi: 10.1007/BF00662396. PMID 8518405
- [Background] Vinceti M, Wei ET, Malagoli C, Bergomi M, Vivoli G. Adverse health effects of selenium in humans. Rev Environ Health. 2001 Jul-Sep;16(4):233-51. doi: 10.1515/reveh.2001.16.4.233. PMID 12041880
- [Background] Youlden DR, Baade PD, Valery PC, Ward LJ, Green AC, Aitken JF. Childhood cancer mortality in Australia. Cancer Epidemiol. 2012 Oct;36(5):476-80. doi: 10.1016/j.canep.2012.06.001. Epub 2012 Jun 26. PMID 22739323
- [Background] Vinceti M, Dennert G, Crespi CM, Zwahlen M, Brinkman M, Zeegers MP, Horneber M, D'Amico R, Del Giovane C. Selenium for preventing cancer. Cochrane Database Syst Rev. 2014 Mar 30;2014(3):CD005195. doi: 10.1002/14651858.CD005195.pub3. PMID 24683040
- [Background] Yang H, Fang J, Jia X, Han C, Chen X, Yang CS, Li N. Chemopreventive effects of early-stage and late-stage supplementation of vitamin E and selenium on esophageal carcinogenesis in rats maintained on a low vitamin E/selenium diet. Carcinogenesis. 2011 Mar;32(3):381-8. doi: 10.1093/carcin/bgq279. Epub 2010 Dec 24. PMID 21186300
- [Background] Zachara BA. Mammalian selenoproteins. J Trace Elem Electrolytes Health Dis. 1992 Sep;6(3):137-51. PMID 1483033
- [Background] Zagrodzki P, Ratajczak R. Selenium status, sex hormones, and thyroid function in young women. J Trace Elem Med Biol. 2008;22(4):296-304. doi: 10.1016/j.jtemb.2008.07.001. Epub 2008 Sep 18. PMID 19013357
- [Background] Zhang S, Li F, Younes M, Liu H, Chen C, Yao Q. Reduced selenium-binding protein 1 in breast cancer correlates with poor survival and resistance to the anti-proliferative effects of selenium. PLoS One. 2013 May 21;8(5):e63702. doi: 10.1371/journal.pone.0063702. Print 2013. PMID 23704933
- See also: Clinical Guidelines for the classification and care of women at risk of familial breast cancer in primary, secondary and tertiary care, NICE, 2013, National Collaborating Centre for Cancer — https://www.nice.org.uk/guidance/cg164/evidence